CLINICAL TRIAL: NCT03741140
Title: Characterizing the Neural Bases of Motivational Disorders After Stroke
Acronym: MOTI-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C17-19; 2018-A00511-54 / 1 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-11-08; First posted 2018-11-14 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Motivation; Apathy; Stroke; Reward; Effort
MeSH Terms: conditions — Stroke; Lethargy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- medial frontal stroke (Other): 20 patients (up to 10 patients can be replaced) with a stroke in the medial frontal lobe will be included in this arm, and will undergo motivation phenotyping.
  Interventions: Diagnostic Test: Motivation tests
- lateral frontal stroke (Other): 20 patients (up to 10 patients can be replaced) with a stroke in the lateral frontal lobe will be included in this arm, and will undergo motivation phenotyping.
  Interventions: Diagnostic Test: Motivation tests
- Healthy participants (Other): 20 healthy participants (up to 10 healthy participants can be replaced) will be included in this arm, and will undergo motivation phenotyping.
  Interventions: Diagnostic Test: Motivation tests

INTERVENTIONS:
Diagnostic Test: Motivation tests — Motivation tests will characterize elementary deficits of motivation

SUMMARY:
The aim of the study is to quantify elementary mechanisms of motivation, with innovative tools adapted to clinical settings, in healthy subjects, and in stroke patients. The secondary aim of the study is to investigate the neural substrates of motivational mechanisms, and to study the impact of lesions in the grey and the white matter, the influence of lesion site.

DETAILED DESCRIPTION:
Disorders of motivation, such as apathy, are among the most prevalent symptoms in neuropsychiatric disorders and during chronic diseases. They have a major impact on patients' physical activity and lifestyle, and on their involvement in their own care. They affect a wide range of morbidity outcomes, alter functional recovery in rehabilitation, impair long-term disability, and prevent patients from returning to an active and independent life. Yet, the neural bases of motivational deficits remain largely unknown. Current diagnostic tools are sparse and cannot distinguish between distinct mechanisms responsible for apathetic syndromes. Besides, current treatments remain extremely limited. However, recent advances in the field of neuroeconomics - the science of decision-making - have provided concept and tools to study the neurobiological bases of elementary cognitive processes underlying motivated behaviors. These theories suggest that the brain implements optimization processes that determine our behaviors by minimizing the cost of our actions while maximizing their expected benefits. The adaptation of tools developed for basic research now enables the assessment of these cognitive mechanisms.

Elementary deficits of motivation will be assessed with a phenotyping battery of motivation tests in 20 healthy subjects (up to 10 healthy subjects can be replaced), 20 patients (up to 10 patients can be replaced) with a stroke in the medial prefrontal cortex, and 20 patients (up to 10 patients can be replaced) with a stroke in the insula. This battery will allow us to characterize, at the patient's level, elementary processes such as the encoding of goal values or effort costs, the modulation of cost with fatigue, and the resolution of cost-benefit trade-offs. Symptom-Lesion mapping studies and voxel-based morphometry studies will be performed using whole brain MRI measures of structural integrity.

ELIGIBILITY:
Inclusion Criteria (healthy volunteers):

* Right-handed
* Age > 18 years old
* Able to squeeze a hand-grip
* Signature of consent form
* Affiliation to an Health Insurance Scheme or beneficiary of such a scheme

Inclusion Criteria (patients):

* Age > 18 years old
* Able to squeeze a hand-grip
* Signature of consent form
* Affiliation to an Health Insurance Scheme or beneficiary of such a scheme
* Stroke of the medial frontal lobe and not affecting the lateral frontal lobe OR stroke of the lateral frontal lobe and not affecting the medial frontal lobe

Exclusion Criteria (healthy volunteers):

* Under justice protection
* History of neurological or psychiatric diseases
* Evolving disease that could impede volunteer participation during the whole study
* Ongoing psychotropic drug or stopped for less than 3 weeks
* Treatment that could interfere with subject performance
* Chronical use of illicit psychoactive drugs or the day of the exam
* Pregnant, parturient or breastfeeding woman
* Exclusion period of another research
* Contra-indication to MRI scan
* Comprehension difficulties or difficulties to perform the study cognitive tests

Exclusion Criteria (patients):

* Under justice protection
* Evolving disease that could impede volunteer participation during the whole study
* Chronical use of illicit psychoactive drugs or the day of the exam
* Pregnant, parturient or breastfeeding woman
* Exclusion period of another research
* Contra-indication to MRI scan
* Comprehension difficulties or difficulties to perform the study cognitive tests
* Brain sequela with important cognitive deficiencies preventing cognitive test interpretation according to the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Reward sensitivity | 1 day
  The reward sensitivity measures the impact of reward values on behavior
Effort sensitivity | 1 day
  The effort sensitivity measures the impact of effort costs on behavior

CONTACTS AND LOCATIONS:
Locations (1):
- Urgences cérébro-vasculaires hopital Pitié-Salpêtrière, Paris, France